CLINICAL TRIAL: NCT05380427
Title: A Phase I Clinical Trial Evaluating the Safety, Tolerability, and Pharmacokinetics of CU-40101 Liniment in Single and Multiple Doses in Adult Male Androgenic Alopecia Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cutia Therapeutics（Wuxi）Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CU-40101-101
Record Dates: First submitted 2022-03-28; First posted 2022-05-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: AGA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Single Dose 1 (Experimental): 0.0025%(0.025 mg/mL)
  Interventions: Drug: CU-40101
- Single Dose 2 (Experimental): 0.005%（于0.05 mg/mL）
  Interventions: Drug: CU-40101
- Single Dose 3 (Experimental): 0.01%（0.1 mg/mL）
  Interventions: Drug: CU-40101
- Single Dose 4 (Experimental): 0.02%（0.2 mg/mL）
  Interventions: Drug: CU-40101
- Multiple Dose 1 (Experimental): 0.05%（0.05 mg/mL）
  Interventions: Drug: CU-40101
- Multiple Dose 2 (Experimental): 0.01%（0.01 mg/mL）
  Interventions: Drug: CU-40101
- Multiple Dose 3 (Experimental): 0.02%（0.02 mg/mL）
  Interventions: Drug: CU-40101
- Placebo (Placebo Comparator): Liniment containing anhydrous ethanol, propylene glycol and polyethylene glycol 400
  Interventions: Drug: CU-40101

INTERVENTIONS:
Drug: CU-40101 — CU-40101，0.0025% CU-40101，0.005% CU-40101，0.01% CU-40101，0.02%

SUMMARY:
1. To evaluate the safety and tolerability of CU-40101 liniment as a single and multiple topical application in adult male androgenic alopecia subjects；
2. To evaluate the pharmacokinetic (PK) characteristics of CU-40101 liniment administered as a single and multiple topical skin application in adult male subjects with androgenic alopecia.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informaed consent.
2. Subject is male, 18-55 years old.
3. Subject has a clinical diagnosis of moderate to severe AGA in temple and vertex region, Ⅲ to Ⅶ on the Modified Norwood-Hamilton Scale.
4. Subject has a body mass index(BMI) of 19 to 28 kg/㎡ inclusive and body weight not less than 50kg.
5. According to the history, physical examination, vital signs, 12-lead electrocardiogram and laboratory examination results, the patient was in good health with no clinically significant abnormalities
6. Subjects (including partners) are willing to take effective contraceptive measures voluntarily within 3 months from signing the informed consent to the last dose.

Exclusion Criteria:

1. Allergic to the study drug or any ingredient in the study drug
2. Skin damage or abnormality at the administration site may affect drug absorption or evaluation, such as dermatitis, scar, tattoo, sunburn, etc
3. Subjects who currently have thyroid disease (including hyperthyroidism, hypothyroidism, etc.) or are currently receiving thyroxine replacement therapy. Thyroid function abnormalities on blood tests at the screening stage or thyroid ultrasound that the investigator judged to be clinically significant must be excluded
4. Any surgical procedures performed within 3 months prior to screening, or planned during the study and within 1 month after the subject completed all study visits
5. A history of clinically significant heart, liver, neurological, respiratory, hematological, digestive, immune, renal, or psychiatric disorders that the investigator believes may confound study results or affect drug absorption, distribution, metabolism, and excretion or place the subject at inappropriate risk

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
AE and SAE | Single dose 29 days; Multiple dose 39 days
  TEAE and SAE will be summarized by dose grouping based on systematic organ Classification (SOC), preferred term (PT) and severity, as well as their relationship to the study drug. Subjects who reported multiple adverse events within the same SOC and PT could only be counted once, according to the highest severity level.
Vital signs | Single dose 29 days; Multiple dose 39 days
  Descriptive statistics summarizing changes in heart rate will be compared between baseline levels at each predetermined point in time.
Vital signs | Single dose 29 days; Multiple dose 39 days
  Descriptive statistics summarizing changes in sitting blood pressure (systolic and diastolic) will be compared between baseline levels at each predetermined point in time.
Vital signs | Single dose 29 days; Multiple dose 39 days
  Descriptive statistics summarizing changes in body temperature will be compared between baseline levels at each predetermined point in time.
12-lead ECG | Single dose 29 days; Multiple dose 39 days
  The number of results of heart rate, QT, QTcF and PR interval will be collected.
  Descriptive statistics summarizing changes of parameters above will be compared between baseline levels at each predetermined point in time.
Laboratory inspection | Single dose 29 days; Multiple dose 39 days
  The number of results of blood routine examination, Blood Biochemical and routine urine examination will be collected Descriptive statistics summarizing changes of parameters above will be compared with baseline levels at each predetermined point in time.
Vital signs | Single dose 29 days; Multiple dose 39 days
  Descriptive statistics summarizing changes in respiration will be compared between baseline levels at each predetermined point in time.
Assessment of topical skin tolerance | Single dose 29 days; Multiple dose 39 days
  The number of erythema, burning/tingling, dryness, pruritus, desquamation of skin and hyperpigmentation after dosing.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Zhejiang, Hangzhou, China